CLINICAL TRIAL: NCT01877668
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Of The Efficacy And Safety Of 2 Doses Of Tofacitinib (CP-690,550) Or Adalimumab In Subjects With Active Psoriatic Arthritis
Brief Title: Efficacy And Safety Of Tofacitinib In Psoriatic Arthritis: Comparator Study
Acronym: OPAL BROADEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921091; 2011-003668-55 (EudraCT Number)
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Psoriatic Arthritis
Keywords: psoriatic arthritis; radiographic changes; active comparator; tofacitinib
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — tofacitinib; BID protein, human; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Tofacitinib 5 mgBID x 12 months (Experimental)
  Interventions: Drug: Tofacitinib 5 mg BID
- Tofacitinib 10 mg BID x 12 months (Experimental)
  Interventions: Drug: Tofacitinib 10 mg BID
- Adalimumab 40 mg q2 weeks x 12 months (Active Comparator)
  Interventions: Drug: Adalimumab
- Placebo x3 months, then tofacitinib 5 mg BIDx 9 months (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo x 3 months, then tofacitinib 10 mg BID x 9 months (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tofacitinib 5 mg BID — Tofacitinib orally (po) 1 tablet of 5 mg and placebo po 1 tablet BID x 12 months Placebo injections subcu every 2 weeks x 12 months
  Arms: Tofacitinib 5 mgBID x 12 months
Drug: Tofacitinib 10 mg BID — Tofacitinib po 2 tablets of 5 mg BID x 12 months Placebo injections subcu every 2 weeks x 12 months
  Arms: Tofacitinib 10 mg BID x 12 months
Drug: Adalimumab — Placebo po 2 tablets BIDx 12 months Adalimumab 40 mg subcu injections every 2 weeks x 12 months
  Arms: Adalimumab 40 mg q2 weeks x 12 months
Drug: Placebo — Placebo po 2 tablets BIDx 3 months followed by tofacitinib po 1 tablet of 5 mg and placebo po 1 tablet BID x 9 months Placebo injections every 2 weeks x 12 months
  Arms: Placebo x3 months, then tofacitinib 5 mg BIDx 9 months
Drug: Placebo — Placebo po 2 tablets BIDx 3 months followed by tofacitinib po 2 tablets (5 mg) BID x 9 months Placebo injections every 2 weeks x 12 months
  Arms: Placebo x 3 months, then tofacitinib 10 mg BID x 9 months

SUMMARY:
This is a 12-month study investigating the effectiveness and safety of tofactinib in treating the signs and symptoms of active psoriatic arthritis and improving physical function and preserving bone structure in patients with an inadequate response to a traditional, nonbiologic disease-modifying antirheumatic drug. Adalimumab is used as a comparator.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged >= 18 years at time of consent.
* Have a diagnosis of Psoriatic arthritis (PsA) of >= 6 months
* Meet the Classification Criteria of PsA (CASPAR) at time of screening
* Must not have been adequately treated with a a traditional non-biologic disease modifying anti-rheumatic drug (DMARD).
* Concurrent treatment with methotrexate, leflunomide, or sulfasalazine allowed and required
* Must not have taken a biologic Tumour Necrosis Factor Inhibitor
* Must have 3 or more swollen joints AND 3 or more tender joints
* Must have active psoriasis skin lesions

Exclusion Criteria:

* Have non-plaque forms of psoriasis, eg erythrodermic, guttate or pustular, with the exception of nail psoriasis which is allowed
* Pregnant or breast feeding, females of child-bearing potential not using highly effective contraception
* New York Heart Association Class III and IV congestive heart failure
* History of hypersensitivity or infusion reaction to biologic agents
* Infection with HIV, hepatitis B virus, hepatitis C virus, or other chronic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2015-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (123):
- United States (24):
  - Rheumatology Associates, PC, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Arizona Arthritis & Rheumatology Associates, P.C., Glendale, Arizona
  - Medvin Clinical Research, Covina, California
  - Desert Medical Advances, Palm Desert, California
  - Advances In Medicine (X-Rays), Rancho Mirage, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Millennium Research, Ormond Beach, Florida
  - Arthritis Center, Inc., Palm Harbor, Florida
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - St. Paul Rheumatology, PA, Eagan, Minnesota
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center (DHMC), Lebanon, New Hampshire
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Drug Shipment/Storage: Huntsman Cancer Hospital at the University of Utah, Salt Lake City, Utah
  - University of Utah Hospital & Clinics, Salt Lake City, Utah
  - Dynacare Laboratories (Specimen processing for shipment), Seattle, Washington
  - Investigational Drug Service Pharmacy, Swedish Medical Center., Seattle, Washington
  - Seattle Rheumatology Associates, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- Australia (6):
  - Rheumatology Research Unit, Maroochydore, Queensland
  - Pacific Private Clinic, Southport, Queensland
  - Monash Health, Monash Medical Centre, Clayton, Victoria
  - Pharmacy Clinical Trials, Clayton, Victoria
  - St. Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - Emeritus Research Pty Ltd, Malvern East, Victoria
- Belgium (2):
  - Hopital Erasme - Clinique Universitaire de Bruxelles, Brussels
  - University Hospital Leuven, Department of Rheumatology, Leuven
- Bulgaria (5):
  - UMHAT "Dr. G. Stranski" EAD, Pleven
  - MHAT"Plovdiv" AD, Plovdiv
  - MHAT "Kaspela" EOOD, Plovdiv
  - UMHAT "Sv. Ivan Rilski" EAD, Sofia
  - MC "New rehabilitation center" EOOD, Rheumatology Cabinet, Stara Zagora
- Canada (3):
  - Rheumatology Research Associates, Edmonton, Alberta
  - K. Papp Clinical Research, Waterloo, Ontario
  - West Island Rheumatology Research Associates, Pointe-Claire, Quebec
- Czechia (13):
  - Revmacentrum MUDr. Mostera, s.r.o., Brno, Czech Republic
  - Revmatologicky Ustav - Lekarna (pharmacy only), Prague, Czech Republic
  - Revmatologicka ambulance, Prague, Czech Republic
  - MEDIGAP, s.r.o. (radiology only), Praha 1 - Nove Mesto, Czech Republic
  - Lekarna Na Lidicke (Pharmacy only), Brno
  - X-MEDICA s.r.o (radiology only), Brno
  - Revmatologie s.r.o., Brno
  - Stavovska s.r.o. (pharmacy only), Brno
  - Vesalion s.r.o., Ostrava
  - Revmatologicky ustav - Lekarna, Prague
  - Revmatologicky ustav, Prague
  - MEDIGAP, s.r.o, Praha 1- Nove Mesto
  - Medical Plus s.r.o. Lekarna Hradebni s. r.o, Uherské Hradiště
- Centre Hospitalier Sud-Francilien - Secretariat de Rhumatologie, Corbeil-Essonnes, France
- Germany (5):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Rheumapraxis Steglitz, Berlin
  - University Hospital of Cologne, Cologne
  - Klinische Forschung Schwerin GmbH, Schwerin
- Hungary (5):
  - Revita Reumatologiai Rendelo, Budapest
  - Qualiclinic Kft., Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont,Reumatologiai osztaly, Budapest
  - Csolnoky Ferenc Korhaz, Radiologiai Osztaly X-Ray Only, Veszprém
  - Csolnoky Ferenc Korhaz, Reumatologiai Osztaly, Veszprém
- Mexico (13):
  - Centro Integral en Reumatologia SA de CV, Guadalajara, Jalisco
  - Centro de Investigacion de Tratamientos Innovadores de Sinaloa, S.C., Culiacán, Sinaloa
  - Laboratorios de Analisis Clinicos CEMSI, Culiacán, Sinaloa
  - Sanatorio CEMSI Chapultepec (For Emergencies Only), Culiacán, Sinaloa
  - Hospital General de Culiacán Dr. Bernardo J. Gastélum, Culiacán, Sinaloa
  - Instituto Medico Panamericano, S.A. de C.V. (For Emergencies Only), Mérida, Yucatán
  - Unidad Reumatologica Las Americas, S.C.P., Mérida, Yucatán
  - Centro de Investigacion Clinica Pensiones, Mérida, Yucatán
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatan, Mérida, Yucatán
  - Hospital Star Medica Merida (For Emergencies Only), Mérida, Yucatán
  - HOSPITAL STAR MEDICA S.A DE C.V- (emergencies only), Mérida, Yucatán
  - Investigacion y Biomedicina de Chihuahua SC, Chihuahua City
  - Cliditer, S. A. de C. V, Mexico City
- Poland (17):
  - Niepubliczny Zaklad Opieki Zdrowotnej Przychodnia Chirurgiczna dla Dzieci "PriamaMed" Sp.P.,", Bialystok
  - ZDROWIE OSTEO-MEDIC s.c. L. i A. Racewicz, A. i J. Supronik, Bialystok
  - ClinicMed Badurski i wspolnicy Spolka Jawna, Bialystok
  - Szpital Uniwersytecki nr 2 im. dr Jana Biziela w Bydgoszczy,, Bydgoszcz
  - Centrum Kliniczno-Badawcze J.Brzezicki, B.Gornikiewicz-Brzezicka Lekarze Spolka Partnerska, Elblag
  - Centrum Radiologii for X-Ray only, Elblag
  - NZOZ Centrum Reumatologiczne Indywidualna Specjalistyczna Praktyka Lekarska Lek. Med. Barbara Bazela, Elblag
  - Przychodnia Specjalistyczna Lekarskiej Spoldzielni Pracy "Medica", Grodzisk Mazowiecki
  - Zespol Poradni Specjalistycznych Reumed Filia Onyksowa, Lublin
  - NZOZ Lecznica MAK-MED S.C., Nadarzyn
  - Prywatna Praktyka Lekarska Prof. UM dr hab. Pawel Hrycaj, Poznan
  - NZOZ Nasz Lekarz Praktyka Grupowa Lekarzy Rodzinnych z Przychodnia Specjalistyczna w Toruniu, Torun
  - Medica Pro Familia Sp. z o.o. S.K.A., Warsaw
  - Rheuma Medicus Zaklad Opieki Zdrowotnej, Warsaw
  - Reumatika Centrum Reumatologii, Warsaw
  - Klinika Ambroziak Estederm Sp. z o.o. ,S.K.A, Warsaw
  - Synexus Polska Sp. z o.o. Oddz. we Wroclawiu, Wroclaw
- Russia (8):
  - Regional State Budgetary Healthcare Institution of Karelia Republic, Petrozavodsk, Karelia Republic
  - State Budgetary Institution of Healthcare of Moscow City Clinical Hospital, Moscow
  - OOO City Neurological Centre "Sibneiromed", Novosibirsk
  - Limited Liability Company Consultative Diagnostic Rheumatology Center "Healthy Joints", Novosibirsk
  - State Institution of Healthcare "Regional Clinical Hospital", Saratov
  - State Budget Educational Institution of Highest Professional Education, Tomsk
  - State Healthcare Institution of Yaroslavl Region Clinical Emergency Hospital n.a. N.V. Solovyev, Yaroslavl
  - State Institution of Healthcare of Yaroslavl Region, Yaroslavl
- Slovakia (4):
  - ROMJAN s.r.o., Reumatologicka ambulancia, Bratislava, Slovak Republic
  - MEDMAN s.r.o. - reumatologicka ambulancia, Martin, Slovak Republic
  - Nestatna reumatologicka ambulancia, Bratislava
  - Reumex s.r.o, Rimavská Sobota
- Spain (6):
  - Hospital Clinico de Santiago, Santiago de Compostela, A Coruna
  - Corporació Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Complexo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Infanta Luisa, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- Taiwan (4):
  - Taipei Veterans General Hospital, Taipei, Taiwan Roc
  - Buddhist Dalin Tzu Chi General Hospital, Chiayi City
  - Chang Gung Medical Foundation-Kaohsiung Branch, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
- United Kingdom (7):
  - Barking Havering and Redbridge University Hospital NHS Trust-King George Hospital, Goodmayes, Essex
  - Barking, Havering and Redbridge University Hospitals NHS Trust, Romford, Essex
  - The Dudley Group NHS Foundation Trust, Dudley, West Midlands
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford, West Yorkshire
  - Bradford Royal Infirmary, BTHFT, Bradford, West Yorkshire
  - Wirral University Teaching Hospital NHS Foundation Trust, Upton, Wirral
  - York Teaching Hospital NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Gossec L, Sellas A, Gruben DC, Valderrama M, Gomez S, Kinch C, Citera G. Response to Tofacitinib in Patients with Psoriatic Arthritis and Probable Anxiety/Depressive Disorder: A Post Hoc Analysis of Phase 3 Trials. Rheumatol Ther. 2025 Dec;12(6):1175-1186. doi: 10.1007/s40744-025-00800-7. Epub 2025 Oct 28. PMID 41148555
- [Derived] Gladman DD, Dougados M, Marzo-Ortega H, Cadatal MJ, Agarwal E, Kinch CD, Nash P. Long-term tofacitinib efficacy and safety in psoriatic arthritis with or without prior biologic DMARD exposure: a post hoc analysis. Rheumatol Adv Pract. 2025 Jan 21;9(2):rkaf008. doi: 10.1093/rap/rkaf008. eCollection 2025. PMID 40241921
- [Derived] Gladman DD, Nash P, Mease PJ, FitzGerald O, Duench S, Cadatal MJ, Masri KR. Efficacy and safety of tofacitinib in an open-label, long-term extension study in patients with psoriatic arthritis who received adalimumab or tofacitinib in a Phase 3 randomized controlled study: a post hoc analysis. Arthritis Res Ther. 2024 Dec 19;26(1):218. doi: 10.1186/s13075-024-03442-2. PMID 39702318
- [Derived] Mease PJ, Orbai AM, FitzGerald O, Bedaiwi M, Dona L Fleishaker, Mundayat R, Young P, Helliwell PS. Efficacy of tofacitinib on enthesitis in patients with active psoriatic arthritis: analysis of pooled data from two phase 3 studies. Arthritis Res Ther. 2023 Aug 22;25(1):153. doi: 10.1186/s13075-023-03108-5. PMID 37608391
- [Derived] Eder L, Gladman DD, Mease P, Pollock RA, Luna R, Aydin SZ, Ogdie A, Polachek A, Gruben D, Cadatal MJ, Kinch C, Strand V. Sex differences in the efficacy, safety and persistence of patients with psoriatic arthritis treated with tofacitinib: a post-hoc analysis of phase 3 trials and long-term extension. RMD Open. 2023 Mar;9(1):e002718. doi: 10.1136/rmdopen-2022-002718. PMID 36958766
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Dougados M, Taylor PC, Bingham CO 3rd, Fallon L, Brault Y, Roychoudhury S, Wang L, Kessouri M. The effect of tofacitinib on residual pain in patients with rheumatoid arthritis and psoriatic arthritis. RMD Open. 2022 Sep;8(2):e002478. doi: 10.1136/rmdopen-2022-002478. PMID 36814062
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Schneeberger EE, Citera G, Nash P, Smolen JS, Mease PJ, Soriano ER, Helling C, Szumski AE, Mundayat R, de Leon DP. Comparison of disease activity index for psoriatic arthritis (DAPSA) and minimal disease activity (MDA) targets for patients with psoriatic arthritis: A post hoc analysis of data from phase 3 tofacitinib studies. Semin Arthritis Rheum. 2023 Feb;58:152134. doi: 10.1016/j.semarthrit.2022.152134. Epub 2022 Nov 13. PMID 36476498
- [Derived] de Vlam K, Mease PJ, Bushmakin AG, Fleischmann R, Ogdie A, Azevedo VF, Merola JF, Woolcott J, Cappelleri JC, Fallon L, Taylor PC. Identifying and Quantifying the Role of Inflammation in Pain Reduction for Patients With Psoriatic Arthritis Treated With Tofacitinib: A Mediation Analysis. Rheumatol Ther. 2022 Oct;9(5):1451-1464. doi: 10.1007/s40744-022-00482-5. Epub 2022 Sep 8. PMID 36076054
- [Derived] Orbai AM, Mease PJ, Helliwell PS, FitzGerald O, Fleishaker DL, Mundayat R, Young P. Effect of tofacitinib on dactylitis and patient-reported outcomes in patients with active psoriatic arthritis: post-hoc analysis of phase III studies. BMC Rheumatol. 2022 Sep 1;6(1):68. doi: 10.1186/s41927-022-00298-4. PMID 36045453
- [Derived] Taylor PC, Bushmakin AG, Cappelleri JC, Young P, Germino R, Merola JF, Yosipovitch G. Relationships of dermatologic symptoms and quality of life in patients with psoriatic arthritis: analysis of two tofacitinib phase III studies. J Dermatolog Treat. 2022 Aug;33(5):2614-2620. doi: 10.1080/09546634.2022.2060924. Epub 2022 Apr 11. PMID 35385361
- [Derived] Gladman DD, Coates LC, Wu J, Fallon L, Bacci ED, Cappelleri JC, Bushmakin AG, Helliwell PS. Time to response for clinical and patient-reported outcomes in patients with psoriatic arthritis treated with tofacitinib, adalimumab, or placebo. Arthritis Res Ther. 2022 Feb 9;24(1):40. doi: 10.1186/s13075-022-02721-0. PMID 35139908
- [Derived] Dikranian A, Gold D, Bessette L, Nash P, Azevedo VF, Wang L, Woolcott J, Shapiro AB, Szumski A, Fleishaker D, Wollenhaupt J. Frequency and Duration of Early Non-serious Adverse Events in Patients with Rheumatoid Arthritis and Psoriatic Arthritis Treated with Tofacitinib. Rheumatol Ther. 2022 Apr;9(2):411-433. doi: 10.1007/s40744-021-00405-w. Epub 2021 Dec 17. PMID 34921355
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Kivitz AJ, FitzGerald O, Nash P, Pang S, Azevedo VF, Wang C, Takiya L. Efficacy and safety of tofacitinib by background methotrexate dose in psoriatic arthritis: post hoc exploratory analysis from two phase III trials. Clin Rheumatol. 2022 Feb;41(2):499-511. doi: 10.1007/s10067-021-05894-2. Epub 2021 Sep 12. PMID 34510295
- [Derived] de Vlam K, Ogdie A, Bushmakin AG, Cappelleri JC, Fleischmann R, Taylor PC, Azevedo V, Fallon L, Woolcott J, Mease PJ. Median time to pain improvement and the impact of baseline pain severity on pain response in patients with psoriatic arthritis treated with tofacitinib. RMD Open. 2021 Jul;7(2):e001609. doi: 10.1136/rmdopen-2021-001609. PMID 34226183
- [Derived] Coates LC, Bushmakin AG, FitzGerald O, Gladman DD, Fallon L, Cappelleri JC, Hsu MA, Helliwell PS. Relationships between psoriatic arthritis composite measures of disease activity with patient-reported outcomes in phase 3 studies of tofacitinib. Arthritis Res Ther. 2021 Mar 26;23(1):94. doi: 10.1186/s13075-021-02474-2. PMID 33766074
- [Derived] Ritchlin CT, Giles JT, Ogdie A, Gomez-Reino JJ, Helliwell P, Young P, Wang C, Wu J, Romero AB, Woolcott J, Stockert L. Tofacitinib in Patients With Psoriatic Arthritis and Metabolic Syndrome: A Post hoc Analysis of Phase 3 Studies. ACR Open Rheumatol. 2020 Oct;2(10):543-554. doi: 10.1002/acr2.11166. Epub 2020 Sep 10. PMID 32910531
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Burmester GR, Curtis JR, Yun H, FitzGerald O, Winthrop KL, Azevedo VF, Rigby WFC, Kanik KS, Wang C, Biswas P, Jones T, Palmetto N, Hendrikx T, Menon S, Rojo R. An Integrated Analysis of the Safety of Tofacitinib in Psoriatic Arthritis across Phase III and Long-Term Extension Studies with Comparison to Real-World Observational Data. Drug Saf. 2020 Apr;43(4):379-392. doi: 10.1007/s40264-020-00904-9. PMID 32006348
- [Derived] Gladman DD, Charles-Schoeman C, McInnes IB, Veale DJ, Thiers B, Nurmohamed M, Graham D, Wang C, Jones T, Wolk R, DeMasi R. Changes in Lipid Levels and Incidence of Cardiovascular Events Following Tofacitinib Treatment in Patients With Psoriatic Arthritis: A Pooled Analysis Across Phase III and Long-Term Extension Studies. Arthritis Care Res (Hoboken). 2019 Oct;71(10):1387-1395. doi: 10.1002/acr.23930. PMID 31112005
- [Derived] Cella D, Wilson H, Shalhoub H, Revicki DA, Cappelleri JC, Bushmakin AG, Kudlacz E, Hsu MA. Content validity and psychometric evaluation of Functional Assessment of Chronic Illness Therapy-Fatigue in patients with psoriatic arthritis. J Patient Rep Outcomes. 2019 May 20;3(1):30. doi: 10.1186/s41687-019-0115-4. PMID 31111255
- [Derived] van der Heijde D, Gladman DD, FitzGerald O, Kavanaugh A, Graham D, Wang C, Fallon L. Radiographic Progression According to Baseline C-reactive Protein Levels and Other Risk Factors in Psoriatic Arthritis Treated with Tofacitinib or Adalimumab. J Rheumatol. 2019 Sep;46(9):1089-1096. doi: 10.3899/jrheum.180971. Epub 2019 Mar 1. PMID 30824647
- [Derived] Strand V, de Vlam K, Covarrubias-Cobos JA, Mease PJ, Gladman DD, Graham D, Wang C, Cappelleri JC, Hendrikx T, Hsu MA. Tofacitinib or adalimumab versus placebo: patient-reported outcomes from OPAL Broaden-a phase III study of active psoriatic arthritis in patients with an inadequate response to conventional synthetic disease-modifying antirheumatic drugs. RMD Open. 2019 Jan 11;5(1):e000806. doi: 10.1136/rmdopen-2018-000806. eCollection 2019. PMID 30713721
- [Derived] Cella D, Wilson H, Shalhoub H, Revicki DA, Cappelleri JC, Bushmakin AG, Kudlacz E, Hsu MA. Content validity and psychometric evaluation of Functional Assessment of Chronic Illness Therapy-Fatigue in patients with psoriatic arthritis. J Patient Rep Outcomes. 2019 Jan 24;3(1):5. doi: 10.1186/s41687-019-0094-5. PMID 30680661 (Retraction: PMID 31139969 J Patient Rep Outcomes. 2019 May 28;3(1):32)
- [Derived] Nash P, Coates LC, Fleischmann R, Papp KA, Gomez-Reino JJ, Kanik KS, Wang C, Wu J, Menon S, Hendrikx T, Ports WC. Efficacy of Tofacitinib for the Treatment of Psoriatic Arthritis: Pooled Analysis of Two Phase 3 Studies. Rheumatol Ther. 2018 Dec;5(2):567-582. doi: 10.1007/s40744-018-0131-5. Epub 2018 Nov 9. PMID 30414064
- [Derived] Helliwell P, Coates LC, FitzGerald O, Nash P, Soriano ER, Elaine Husni M, Hsu MA, Kanik KS, Hendrikx T, Wu J, Kudlacz E. Disease-specific composite measures for psoriatic arthritis are highly responsive to a Janus kinase inhibitor treatment that targets multiple domains of disease. Arthritis Res Ther. 2018 Oct 29;20(1):242. doi: 10.1186/s13075-018-1739-0. PMID 30373651
- [Derived] Mease P, Hall S, FitzGerald O, van der Heijde D, Merola JF, Avila-Zapata F, Cieslak D, Graham D, Wang C, Menon S, Hendrikx T, Kanik KS. Tofacitinib or Adalimumab versus Placebo for Psoriatic Arthritis. N Engl J Med. 2017 Oct 19;377(16):1537-1550. doi: 10.1056/NEJMoa1615975. PMID 29045212
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921091&StudyName=Efficacy%20And%20Safety%20Of%20Tofacitinib%20In%20Psoriatic%20Arthritis%3A%20Comparator%20Study

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 611 participants screened for entry into the study, 422 received treatment.
Groups:
- Tofacitinib, 5 mg, Twice Daily: Participants received 1 tofacitinib 5-mg tablet twice daily, 1 placebo tablet twice daily, and subcutaneous placebo administered every 2 weeks.
- Tofacitinib, 10 mg, Twice Daily: Participants received 2 tofacitinib 5-mg tablets twice daily and subcutaneous placebo every 2 weeks.
- Adalimumab, 40 mg, Every 2 Weeks: Participants received 2 placebo tablets twice daily and adalimumab, 40 mg, administered subcutaneously every 2 weeks.
- Placebo/Tofacitinib, 5 mg, Twice Daily: Participants received 2 placebo tablets twice daily and subcutaneous placebo every 2 weeks for 3 months. At the end of this period, participants received 1 tofacitinib 5-mg tablet twice daily, 1 placebo tablet twice daily, and subcutaneous placebo every 2 weeks.
- Placebo/Tofacitinib, 10 mg, Twice Daily: Participants received 2 placebo tablets twice daily and subcutaneous placebo every 2 weeks for 3 months. At the end of this period, participants received 2 tofacitinib 5-mg tablets twice daily and subcutaneous placebo every 2 weeks.
Period: Overall Study
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily
Started | 107 (Received treatment) | 104 (Received treatment) | 106 (Received treatment) | 52 (Received treatment) | 53 (Received treatment)
Completed | 96 | 96 | 94 | 44 | 43
Not Completed | 11 | 8 | 12 | 8 | 10
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — No longer met study criteria | 1 | 0 | 1 | 0 | 0
Not completed — Insufficient clinical response | 0 | 1 | 2 | 2 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 3 | 2 | 2
Not completed — Other | 1 | 1 | 1 | 1 | 3
Not completed — Protocol Violation | 1 | 1 | 0 | 0 | 3
Not completed — Adverse event related to study drug | 2 | 2 | 2 | 2 | 1
Not completed — Adverse event unrelated to study drug | 4 | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Total
Number analyzed (Participants) | 107 | 104 | 106 | 52 | 53 | 422
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.4 (12.6) | 46.9 (12.4) | 47.4 (11.3) | 46.1 (10.4) | 49.3 (13.8) | 47.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 62 | 50 | 28 | 28 | 225
  Male | 50 | 42 | 56 | 24 | 25 | 197

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting American College of Rheumatology Response Criteria ≥20% (ACR20): Month 3
Description: ACR20 was calculated as a ≥20% improvement from baseline in tender/painful and swollen joint counts and ≥20% improvement from baseline in 3 of the 5 remaining ACR core set measures: patient's global assessment of arthritis, physician's global assessment of arthritis, patient's assessment of arthritis pain, health assessment questionnaire - disability index (HAQ-DI), and C-reactive protein (CRP).
Time Frame: At end of Month 3
Population: All participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: Percentage or participants
Groups:
- Placebo: Participants received 2 placebo tablets twice daily and subcutaneous placebo every 2 weeks for 3 months.
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo
Number analyzed (Participants) | 107 | 104 | 106 | 105
Percentage or participants | 50.47 | 60.58 | 51.89 | 33.33
Statistical Analysis 1: Comparison: Tofacitinib, 5 mg, Twice Daily vs Placebo; Test type: Superiority or Other; p = 0.0102, Large sample approximation; Missing response (MR)=non-response (NR); Risk Difference (RD) = 17.13, 95% CI 2-sided [4.06 to 30.21], Standard Error of Mean 6.67
Statistical Analysis 2: Comparison: Tofacitinib, 10 mg, Twice Daily vs Placebo; Test type: Superiority or Other; p < 0.0001, Large sample approximation; MR=NR; Risk Difference (RD) = 27.24, 95% CI 2-sided [14.22 to 40.26], Standard Error of Mean 6.64
Statistical Analysis 3: Comparison: Adalimumab, 40 mg, Every 2 Weeks vs Placebo; Test type: Superiority or Other; p = 0.0055, Large sample approximation; MR=NR; Risk Difference (RD) = 18.55, 95% CI 2-sided [5.45 to 31.66], Standard Error of Mean 6.69

2. Primary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score
Description: The HAQ-DI assesses the difficulty a participant has had in the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2-3 items. For each question, level of difficulty is scored from 0 to 3 with 0=no difficulty, 1=some difficulty, 2=much difficulty, and 3=unable to do. The score for each domain is the maximum (worst) score from the items/questions within the domain. Higher score indicates greater disability.
Time Frame: From Baseline to Month 3
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo
Number analyzed (Participants) | 107 | 104 | 106 | 104
Units on a scale | -0.3499 (0.04665) | -0.3998 (0.04716) | -0.3808 (0.04767) | -0.1802 (0.05031)
Statistical Analysis 1: Comparison: Tofacitinib, 5 mg, Twice Daily vs Placebo; Test type: Superiority or Other; p = 0.0062, Mixed Models Analysis; No imputation; Mean Difference (Net) = -0.1697, 95% CI 2-sided [-0.2910 to -0.0483], Standard Error of Mean 0.06173
Statistical Analysis 2: Comparison: Tofacitinib, 10 mg, Twice Daily vs Placebo; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; No imputation; Mean Difference (Net) = -0.2196, 95% CI 2-sided [-0.3411 to -0.0980], Standard Error of Mean 0.06184
Statistical Analysis 3: Comparison: Adalimumab, 40 mg, Every 2 Weeks vs Placebo; Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis; No imputation; Mean Difference (Net) = -0.2005, 95% CI 2-sided [-0.3213 to -0.0797], Standard Error of Mean 0.06145

3. Secondary Outcome: Change From Baseline in the Van Der Heijdel Modified Total Sharp Score (mTSS) for Psoriatic Arthritis
Description: Assessment of joint damage includes a joint erosion score (range 0-320) and a joint space narrowing (JSN) score (range 0-208). The mTSS is the sum of the erosion and JSN scores (range 0-528). A higher score indicates more severe disease status. If a component score is missing, the mTSS will be missing.
Time Frame: From Baseline to Month 12
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Placebo/Tofacitinib, 5 mg, Twice Daily; Placebo/Tofacitinib, 10 mg, Twice Daily: Participants received 2 placebo tablets twice daily and subcutaneous placebo every 2 weeks for 3 months. At the end of this period, participants received 2 tofacitinib 5-mg tablets twice daily and subcutaneous placebo every 2 weeks.
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily
Number analyzed (Participants) | 98 | 99 | 95 | 48 | 45
Units on a scale | 0.01 (0.067) | -0.01 (0.067) | -0.07 (0.069) | 0.00 (0.094) | 0.09 (0.099)

4. Secondary Outcome: Percentage of Participants With Progressed Modified Total Sharp Score (mTSS) at Month 12
Description: Assessment of joint damage includes a joint erosion score (range 0-320) and a JSN score (range 0-208). The mTSS is the sum of the erosion and JSN scores (range 0-528). A higher score indicates more severe disease status. If a component score is missing, the mTSS will be missing. Progressor is defined as an increase in mTSS >0.5 from baseline.
Time Frame: At Month 12
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily
Number analyzed (Participants) | 98 | 99 | 95 | 48 | 45
Percentage of participants | 4.08 | 5.05 | 2.11 | 4.17 | 8.89

5. Secondary Outcome: Percentage of Participants Meeting American College of Rheumatology Response Criteria ≥50% (ACR50) at Week 2 and Months 1, 2, 3, 4, 6, 9, and 12
Description: ACR50 was calculated as a ≥50% improvement from baseline in tender/painful and swollen joint counts and ≥50% improvement from baseline in 3 of the 5 remaining ACR core set measures: patient's global assessment of arthritis, physician's global assessment of arthritis, patient's assessment of arthritis pain, HAQ-DI, and CRP.
Time Frame: At Week 2 and Months 1, 2, 3, 4, 6, 9, and 12
Population: All participants who were randomized and received at least 1 dose of study drug. n=number of responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 107 | 104 | 106 | 52 | 53 | 105
Percentage of participants
  Week 2 (n=7, 7, 5, NA, NA, 1) | 6.54 | 6.73 | 4.72 | NA — Results not reported for this group. | NA — Results not reported for this group. | 0.95
  Month 1 (n=13, 20,12, NA, NA, 5) | 12.15 | 19.23 | 11.32 | NA — Results not reported for this group. | NA — Results not reported for this group. | 4.76
  Month 2 (n=23, 34, 24, NA, NA, 8) | 21.50 | 32.69 | 22.64 | NA — Results not reported for this group. | NA — Results not reported for this group. | 7.62
  Month 3 (n=30, 42, 35, NA, NA, 10) | 28.04 | 40.38 | 33.02 | NA — Results not reported for this group. | NA — Results not reported for this group. | 9.52
  Month 4 (n=38, 39, 34, 11, 17, NA) | 35.51 | 37.50 | 32.08 | 21.15 | 32.08 | NA — Results not reported for this group.
  Month 6 (n=41, 48, 45, 17, 14, NA) | 38.32 | 46.15 | 42.45 | 32.69 | 26.42 | NA — Results not reported for this group.
  Month 9 (n=45, 48, 49, 22, 23, NA) | 42.06 | 46.15 | 46.23 | 42.31 | 43.40 | NA — Results not reported for this group.
  Month 12 (n=48, 50, 43, 21, 19, NA) | 44.86 | 48.08 | 40.57 | 40.38 | 35.85 | NA — Results not reported for this group.

6. Secondary Outcome: Percentage of Participants Meeting American College of Rheumatology Response Criteria ≥70% (ACR70) at Week 2 and Months 1, 2, 3, 4, 6, 9, and 12
Description: ACR70 was calculated as a ≥70% improvement from baseline in tender/painful and swollen joint counts and ≥70% improvement from baseline in 3 of the 5 remaining ACR core set measures: patient's global assessment of arthritis, physician's global assessment of arthritis, patient's assessment of arthritis pain, HAQ-DI, and CRP.
  .
Time Frame: At Week 2 and Months 1, 2, 3, 4, 6, 9, and 12
Population: All participants who were randomized and received at least 1 dose of study drug. n=number of responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 107 | 104 | 106 | 52 | 53 | 105
Percentage of participants
  Week 2 (n=0, 3, 1, NA, NA, 0) | 0.00 | 2.88 | 0.94 | NA — Results not reported for this group. | NA — Results not reported for this group. | 0.00
  Month 1 (n=5, 8, 4, NA, NA, 1) | 4.67 | 7.69 | 3.77 | NA — Results not reported for this group. | NA — Results not reported for this group. | 0.95
  Month 2 (n=10, 14, 13, NA, NA, 2) | 9.35 | 13.46 | 12.26 | NA — Results not reported for this group. | NA — Results not reported for this group. | 1.90
  Month 3 (n=18, 15, 20, NA, NA, 5) | 16.82 | 14.42 | 18.87 | NA — Results not reported for this group. | NA — Results not reported for this group. | 4.76
  Month 4 (n=24, 23, 21, 7, 8, NA) | 22.43 | 22.12 | 19.81 | 13.46 | 15.09 | NA — Results not reported for this group.
  Month 6 (n=19, 33, 32, 10, 7, NA) | 17.76 | 31.73 | 30.19 | 19.23 | 13.21 | NA — Results not reported for this group.
  Month 9 (n=21, 31, 30, 15, 12, NA) | 19.63 | 29.81 | 28.30 | 28.85 | 22.64 | NA — Results not reported for this group.
  Month 12 (n=25, 32, 31, 12, 12, NA) | 23.36 | 30.77 | 29.25 | 23.08 | 22.64 | NA — Results not reported for this group.

7. Secondary Outcome: Percentage of Participants Meeting American College of Rheumatology Response Criteria ≥20% (ACR20) at Week 2 and Months 1, 2, 4, 6, 9, and 12
Description: ACR20 was calculated as a ≥20% improvement from baseline in tender/painful and swollen joint counts and ≥20% improvement from baseline in 3 of the 5 remaining ACR core set measures: patient's global assessment of arthritis, physician's global assessment of arthritis, patient's assessment of arthritis pain, HAQ-DI, and CRP.
Time Frame: At Week 2 and Months 1, 2, 4, 6, 9, and 12
Population: All participants who were randomized and received at least 1 dose of study drug. n=number of responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 107 | 104 | 106 | 52 | 53 | 105
Percentage of participants
  Week 2 (n=24, 33, 23, NA, NA, 6) | 22.43 | 31.73 | 21.70 | NA — Results not reported for this group. | NA — Results not reported for this group. | 5.71
  Month 1 (n=37, 50, 30, NA, NA, 11) | 34.58 | 48.08 | 28.30 | NA — Results not reported for this group. | NA — Results not reported for this group. | 10.48
  Month 2 (n=47, 57, 62, NA, NA, 28) | 43.93 | 54.81 | 58.49 | NA — Results not reported for this group. | NA — Results not reported for this group. | 26.67
  Month 4 (n=65, 60, 61, 27, 28, NA) | 60.75 | 57.69 | 57.55 | 51.92 | 52.83 | NA — Results not reported for this group.
  Month 6 (n=63, 70, 68, 31, 30, NA) | 58.88 | 67.31 | 64.15 | 59.62 | 56.60 | NA — Results not reported for this group.
  Month 9 (n=73, 76, 73, 35, 37, NA) | 68.22 | 73.08 | 68.87 | 67.31 | 69.81 | NA — Results not reported for this group.
  Month 12 (n=73, 73, 64, 35, 31, NA) | 68.22 | 70.19 | 60.38 | 67.31 | 58.49 | NA — Results not reported for this group.

8. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score
Description: as for outcome 2
Time Frame: From Baseline to Week 2 and Months 1, 2, 4, 6, 9, and 12
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable. n=number of participants evaluable at each visit.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 107 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Week 2 (n=106, 102, 103, NA, NA, 102) | -0.1842 (0.04131) | -0.2089 (0.04208) | -0.2129 (0.04246) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -0.0837 (0.04549)
  Month 1 (n=105, 103, 104, NA, NA, 103) | -0.2048 (0.04363) | -0.2676 (0.04426) | -0.3028 (0.04465) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -0.1224 (0.04755)
  Month 2 (n=104, 104, 104, NA, NA, 102) | -0.2713 (0.04626) | -0.4009 (0.04678) | -0.3736 (0.04719) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -0.1682 (0.04998)
  Month 4 (n=102, 100, 102, 50, 50, NA) | -0.4231 (0.04982) | -0.4407 (0.05039) | -0.3643 (0.05069) | -0.2850 (0.07075) | -0.3302 (0.07128) | NA (NA) — Results were not reported for this group.
  Month 6 (n=100, 100, 99, 48, 48, NA) | -0.4471 (0.05136) | -0.4611 (0.05179) | -0.4259 (0.05227) | -0.3142 (0.07315) | -0.3841 (0.07369) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 96, 96, 47, 45, NA) | -0.5119 (0.05038) | -0.4847 (0.05096) | -0.4304 (0.05143) | -0.3843 (0.07185) | -0.4839 (0.07276) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | -0.5391 (0.05324) | -0.5104 (0.05365) | -0.4478 (0.05426) | -0.4104 (0.07646) | -0.4569 (0.07704) | NA (NA) — Results were not reported for this group.

9. Secondary Outcome: Change From Baseline in American College of Rheumatology Response Criteria Components: C-reactive Protein Levels
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: From Baseline to end of Month 3
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo
Number analyzed (Participants) | 107 | 104 | 106 | 104
mg/L | -5.5981 (0.80656) | -6.6004 (0.80822) | -7.8955 (0.82547) | -0.8643 (0.86304)

10. Secondary Outcome: Change From Baseline in American College of Rheumatology Response Criteria Components Score: Patient's Assessment of Arthritis Pain
Description: Participants assessed the severity of their arthritis pain using a 100-mm visual analog scale (VAS) by placing a mark on the scale between 0 (no pain) and 100 (most severe pain), which corresponded to the magnitude of their pain.
Time Frame: From Baseline to end of Month 3
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo
Number analyzed (Participants) | 107 | 104 | 105 | 104
mm | -21.49 (2.325) | -27.10 (2.342) | -21.87 (2.389) | -10.22 (2.499)

11. Secondary Outcome: Change From Baseline in American College of Rheumatology Response Criteria Components Score: Patient's Global Assessment of Arthritis
Description: Participant answered the following question, "Considering all the ways your arthritis affects you, how are you feeling today?" The participant's response was recorded using a 100 mm VAS by placing a mark on the scale between 0 (very well) and 100 (very poorly).
Time Frame: From Baseline to end of Month 3
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo
Number analyzed (Participants) | 107 | 104 | 106 | 104
mm | -20.08 (2.275) | -25.50 (2.291) | -21.47 (2.328) | -11.40 (2.439)

12. Secondary Outcome: Change From Baseline in American College of Rheumatology Response Criteria Components Score: Physician's Global Assessment of Arthritis
Description: The blinded investigator or qualified assessor assessed how the participant's overall arthritis appeared at the time of the visit. This was an evaluation based on the participant's disease signs, functional capacity and physical examination, and was independent of the Patient's Global Assessment of Arthritis. The investigator's response was recorded using a 100 mm VAS by placing a mark on the scale between 0 (very good) and 100 (very poor).
Time Frame: From Baseline to end of Month 3
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo
Number analyzed (Participants) | 107 | 103 | 106 | 104
mm | -27.44 (1.998) | -33.74 (2.021) | -29.02 (2.043) | -22.26 (2.121)

13. Secondary Outcome: Change From Baseline in American College of Rheumatology Response Criteria Components Score: Swollen Joint Count
Description: Swollen joint counts are considered the most specific quantitative clinical measure used to assess the status of participants with inflammatory types of arthritis. Sixty six (66) joints were assessed by a blinded assessor to determine the number of joints that were considered swelling.
Time Frame: From Baseline to end of Month 3
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Joints
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo
Number analyzed (Participants) | 107 | 104 | 106 | 104
Joints | -6.5 (0.58) | -7.6 (0.58) | -6.5 (0.59) | -4.8 (0.62)

14. Secondary Outcome: Change From Baseline in American College of Rheumatology Response Criteria Components Score: Tender/Painful Joint Count
Description: Tender/painful joint counts are considered the most specific quantitative clinical measure used to assess the status of participants with inflammatory types of arthritis. Sixty eight (68) joints were assessed by a blinded assessor to determine the number of joints that were considered tender or painful.
Time Frame: From Baseline to end of Month 3
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Joints
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo
Number analyzed (Participants) | 107 | 104 | 106 | 104
Joints | -8.7 (1.04) | -11.0 (1.05) | -7.6 (1.07) | -6.9 (1.10)

15. Secondary Outcome: Percentage of Participants Meeting Psoriatic Arthritis Response Criteria (PsARC) at Week 2 and Months 1, 2, 3, 4, 6, 9, and 12
Description: The PsARC covers 4 measures: Tender/painful joint count, swollen joint count, the Physician's Global Assessment of Arthritis, and the Patient's Global Assessment of Arthritis. The PsARC response is defined as improvement in 2 of 4 items, 1 of which must be joint pain or swelling, without worsening in any measure. Improvement criteria: ≥20% improvement in Physician's Global Assessment of Arthritis; ≥20% improvement in Patient's Global Assessment of Arthritis; ≥30% improvement in tender joint count; and ≥30% improvement in swollen joint count.
Time Frame: At Week 2 and Months 1, 2, 3, 4, 6, 9, and 12
Population: All participants who were randomized and received at least 1 dose of study drug. n=number of responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 107 | 104 | 106 | 52 | 53 | 105
Percentage of participants
  Week 2 (n=34, 42, 23, NA, NA, 10) | 31.78 | 40.38 | 21.70 | NA — Results not reported for this group. | NA — Results not reported for this group. | 9.52
  Month 1 (n=45, 51, 43, NA, NA, 23) | 42.06 | 49.04 | 40.57 | NA — Results not reported for this group. | NA — Results not reported for this group. | 21.90
  Month 2 (n=54, 69, 62, NA, NA, 36) | 50.47 | 66.35 | 58.49 | NA — Results not reported for this group. | NA — Results not reported for this group. | 34.29
  Month 3 (n=55, 73, 65, NA, NA, 47) | 51.40 | 70.19 | 61.32 | NA — Results not reported for this group. | NA — Results not reported for this group. | 44.76
  Month 4 (n=68, 68, 71, 32, 30, NA) | 63.55 | 65.38 | 66.98 | 61.54 | 56.60 | NA — Results not reported for this group.
  Month 6 (n=61, 75, 71, 35, 35, NA) | 57.01 | 72.12 | 66.98 | 67.31 | 66.04 | NA — Results not reported for this group.
  Month 9 (n=75, 73, 71, 36, 37, NA) | 70.09 | 70.19 | 66.98 | 69.23 | 69.81 | NA — Results not reported for this group.
  Month 12 (n=69, 76, 69, 39, 33, NA) | 64.49 | 73.08 | 65.09 | 75.00 | 62.26 | NA — Results not reported for this group.

16. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Psoriasis (PGA-PsO) Response
Description: The PGA-PsO is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are rated separately over the whole body according to a 5-point severity scale, scored as 0=none; 1, 2, 3, or 4=most severe. The severity rating scores are summed and the average taken; the total average is rounded to the nearest whole number score to determine a PGA-PsO score on a scale of 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe).
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: All participants who were randomized, received at least 1 dose of study drug with baseline PGA-PsO>0 and were evaluable. n=number of participants evaluable at each visit.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 101 | 98 | 102 | 50 | 50 | 100
Units on a scale
  Month 1 (n=100, 96, 100, NA, NA, 99) | -0.7 (0.07) | -0.8 (0.08) | -0.5 (0.08) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | -0.2 (0.08)
  Month 3 (n=98, 97, 98, NA, NA, 98) | -1.0 (0.08) | -1.2 (0.08) | -1.0 (0.09) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | -0.4 (0.09)
  Month 6 (n=96, 94, 96, 46, 46, NA) | -0.9 (0.09) | -1.3 (0.09) | -1.2 (0.09) | -0.7 (0.12) | -0.9 (0.13) | NA (NA) — Results not reported for this group.
  Month 9 (n=95, 91, 94, 45, 44, NA) | -1.0 (0.09) | -1.5 (0.09) | -1.2 (0.09) | -0.7 (0.12) | -1.3 (0.13) | NA (NA) — Results not reported for this group.
  Month 12 (n=91, 90, 92, 41, 43, NA) | -1.2 (0.09) | -1.5 (0.09) | -1.2 (0.09) | -0.9 (0.13) | -1.3 (0.13) | NA (NA) — Results not reported for this group.

17. Secondary Outcome: Percentage of Participants With Psoriasis Area and Severity Index 75 (PASI75) Response at Months 1, 3, 6, 9, and 12
Description: PASI determines psoriasis severity based on lesion severity & percentage body surface area (BSA) affected. Lesion severity is assessed for erythema, induration, & scaling, evaluated separately for head & neck, upper limbs, trunk, & lower limbs & rated for each body area according to a 5 point scale: 0=no involvement; 1=slight; 2=moderate; 3=marked; 4=very marked. BSA involvement is the extent (%) of body area affected by psoriasis & is assigned a score: 0=no involvement; 1=0-9%; 2=10-29%; 3=30-49%; 4=50-69%; 5=70-89%; 6=90-100%. In each area, sum of severity rating scores is multiplied by the score representing the percentage of area involved by psoriasis, multiplied by a weighting factor (head 0.1; upper limbs 0.2; trunk 0.3; lower limbs 0.4). The sum of numbers obtained for the 4 body areas is the PASI score & can vary in increments of 0.1 & range from 0.0 to 72.0, higher scores represent greater severity of psoriasis. PASI75 is defined as a 75% reduction from baseline in PASI.
Time Frame: At Months 1, 3, 6, 9, and 12
Population: All participants who were randomized and received at least 1 dose of study drug with PASI>0 and BSA ≥3% at baseline. n=number of responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 82 | 70 | 77 | 42 | 40 | 82
Percentage of participants
  Month 1 (n=19, 19, 11, NA, NA, 4) | 23.17 (4.66) | 27.14 (5.32) | 14.29 (3.99) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | 4.88 (2.38)
  Month 3 (n=35, 31, 30, NA, NA, 12) | 42.68 (5.46) | 44.29 (5.94) | 38.96 (5.56) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | 14.63 (3.90)
  Month 6 (n=38, 42, 42, 12, 17, NA) | 46.34 (5.51) | 60.00 (5.86) | 54.55 (5.67) | 28.57 (6.97) | 42.50 (7.82) | NA (NA) — Results not reported for this group.
  Month 9 (n=36, 48, 45, 14, 20, NA) | 43.90 (5.448) | 68.57 (5.55) | 58.44 (5.62) | 33.33 (7.27) | 50.00 (7.91) | NA (NA) — Results not reported for this group.
  Month 12 (n=46, 47, 43, 15, 21, NA) | 56.10 (5.48) | 67.14 (5.61) | 55.84 (5.66) | 35.71 (7.39) | 52.50 (7.90) | NA (NA) — Results not reported for this group.

18. Secondary Outcome: Change From Baseline in Dactylitis Severity Score (DSS)
Description: Dactylitis is characterized by swelling of the entire finger or toe. The DSS is a function of finger circumference and tenderness, assessed and summed across all dactylitic digits. The severity of dactylitis is scored on a scale of 0-3, where 0=no tenderness and 3=extreme tenderness in each digit of the hands and feet. The range of total dactylitis scores for a patient is 0-60. Higher score indicates greater degree of tenderness.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: All participants who were randomized, received at least 1 dose of study drug with baseline DSS>0 and were evaluable. n=number of participants evaluable at each visit.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 60 | 60 | 58 | 29 | 28 | 57
Units on a scale
  Month 1 (n=58, 59, 56, NA, NA, 56) | -1.8 (0.91) | -3.1 (0.87) | -2.1 (0.93) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | 0.6 (1.02)
  Month 3 (n=58, 60 , 56, NA, NA, 55) | -3.5 (0.95) | -5.5 (0.91) | -4.0 (0.97) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | -2.0 (1.06)
  Month 6 (n=58, 59, 55, 28, 25, NA) | -5.2 (1.01) | -6.4 (0.99) | -5.4 (1.03) | -5.9 (1.45) | -5.2 (1.50) | NA (NA) — Results not reported for this group.
  Month 9 (n=57, 59, 53, 27, 25, NA) | -7.0 (0.60) | -7.2 (0.58) | -6.5 (0.63) | -5.3 (0.87) | -7.9 (0.89) | NA (NA) — Results not reported for this group.
  Month 12 (n=54, 58, 52, 26, 24, NA) | -7.4 (0.65) | -7.5 (0.62) | -6.1 (0.67) | -6.7 (0.93) | -7.7 (0.96) | NA (NA) — Results not reported for this group.

19. Secondary Outcome: Change From Baseline in the Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index
Description: The SPARCC Enthesitis Index identifies the presence or absence of tenderness at 16 enthesial sites, including the bilateral Achilles tendons, plantar fascia insertion at the calcaneus, patellar tendon insertion at the base of the patella, quadriceps insertion into the superior border of the patella, supraspinatus insertion into the greater tuberosity of the humerus, and medial and lateral epicondyles. On examination, tenderness is recorded as present (1) or absent (0) for each of the 16 sites, with an overall total score ranging from 0 to 16. Higher score indicates a greater number of sites that are affected by enthesitis.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: All participants who were randomized, received at least 1 dose of study drug with baseline SPARCC Enthesitis Score>0 and were evaluable. n=number of participants evaluable at each visit.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 80 | 81 | 82 | 38 | 41 | 79
Units on a scale
  Month 1 (n=79, 80, 80, NA, NA, 78) | -0.83 (0.317) | -1.27 (0.321) | -0.95 (0.336) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | -0.58 (0.355)
  Month 3 (n=77, 79, 79, NA, NA, 78) | -1.84 (0.363) | -2.41 (0.364) | -1.90 (0.375) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | -1.17 (0.393)
  Month 6 (n=76, 78, 76, 33, 39, NA) | -2.4 (0.34) | -2.6 (0.34) | -2.3 (0.35) | -2.4 (0.50) | -2.5 (0.48) | NA (NA) — Results not reported for this group.
  Month 9 (n=75, 75, 73, 34, 37, NA) | -2.9 (0.31) | -2.6 (0.32) | -3.0 (0.33) | -2.8 (0.46) | -3.2 (0.44) | NA (NA) — Results not reported for this group.
  Month 12 (n=72, 73, 72, 31, 37, NA) | -3.2 (0.33) | -3.1 (0.33) | -2.8 (0.35) | -2.5 (0.49) | -3.2 (0.46) | NA (NA) — Results not reported for this group.

20. Secondary Outcome: Change From Baseline in the Leeds Enthesitis Index (LEI)
Description: Enthesitis is inflammation in the tendon, ligament, and joint capsule fiber insertion into bone. The LEI assesses enthesitis in 6 sites. Tenderness is recorded as either present (1) or absent (0) for each of the 6 sites, for an total score of 0-6. Higher score indicates a greater number of sites that are affected by enthesitis.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: All participants who were randomized, received at least 1 dose of study drug with baseline LEI>0 and were evaluable. n=number of participants evaluable at each visit.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 74 | 64 | 76 | 31 | 34 | 65
Units on a scale
  Month 1 (n=74, 63, 75, NA, NA, 65) | -0.41 (0.192) | -0.57 (0.213) | -0.42 (0.203) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | -0.26 (0.219)
  Month 3 (n=70, 63, 73, NA, NA, 63) | -0.82 (0.221) | -1.46 (0.240) | -1.10 (0.228) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | -0.43 (0.246)
  Month 6 (n=72, 61, 71, 27, 31, NA) | -1.3 (0.21) | -1.2 (0.23) | -1.3 (0.22) | -1.0 (0.32) | -1.3 (0.30) | NA (NA) — Results not reported for this group.
  Month 9 (n=70, 58, 68, 27, 29, NA) | -1.4 (0.20) | -1.3 (0.23) | -1.5 (0.21) | -1.4 (0.31) | -1.7 (0.30) | NA (NA) — Results not reported for this group.
  Month 12 (n=67, 56, 67, 24, 29, NA) | -1.7 (0.19) | -1.6 (0.21) | -1.6 (0.20) | -1.4 (0.30) | -1.9 (0.28) | NA (NA) — Results not reported for this group.

21. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2 (SF-36v2) Acute, Physical Component Summary Score
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. An additional item measures health transition. The 8 health domains are aggregated into two summary scores known as the physical component summary (PCS) score and the mental component summary (MCS) score. Norm-based domain scores, PCS and MCS scores are used in the analyses; each of which has a population mean of 50 with a standard deviation (SD) of 10 points, and ranges from minus infinity to plus infinity. A higher PCS score represents better physical health status.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103,104, NA, NA, 103) | 3.39 (0.638) | 4.66 (0.645) | 4.00 (0.655) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | 1.54 (0.700)
  Month 3 (n=102, 103,100, NA, NA, 102) | 5.51 (0.733) | 5.69 (0.735) | 6.23 (0.748) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | 2.68 (0.785)
  Month 6 (n=100, 100, 98, 48, 48, NA) | 6.72 (0.773) | 6.70 (0.777) | 6.26 (0.788) | 5.86 (1.101) | 6.07 (1.112) | NA (NA) — Results not reported for this group.
  Month 9 (n=99, 97, 95, 47, 46, NA) | 7.52 (0.781) | 7.21 (0.787) | 6.91 (0.798) | 6.16 (1.115) | 7.15 (1.130) | NA (NA) — Results not reported for this group.
  Month 12 (n=96, 96, 94, 44, 43, NA) | 7.61 (0.806) | 7.67 (0.810) | 6.74 (0.822) | 5.82 (1.160) | 5.72 (1.177) | NA (NA) — Results not reported for this group.

22. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2 (SF-36v2), Acute, Mental Component Summary Score
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. An additional item measures health transition. The 8 health domains are aggregated into two summary scores known as the PCS score and the MCS score. Norm-based domain scores, PCS and MCS scores are used in the analyses; each of which has a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher MCS score represents better mental health status.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103,104,NA, NA, 103) | 4.12 (0.841) | 3.63 (0.849) | 2.13 (0.871) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | 3.19 (0.917)
  Month 3 (n=102, 103,100, NA, NA, 102) | 4.35 (0.909) | 4.20 (0.909) | 3.13 (0.938) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | 3.27 (0.976)
  Month 6 (n=100, 100, 98, 48, 48, NA) | 5.70 (0.927) | 5.51 (0.930) | 4.58 (0.955) | 4.50 (1.319) | 3.62 (1.331) | NA (NA) — Results not reported for this group.
  Month 9 (n=99, 97, 95, 47, 46, NA) | 5.07 (0.974) | 6.20 (0.982) | 3.68 (1.005) | 4.61 (1.391) | 6.03 (1.409) | NA (NA) — Results not reported for this group.
  Month 12 (n=96, 96, 94, 44, 43, NA) | 4.82 (1.012) | 6.26 (1.016) | 4.81 (1.039) | 4.51 (1.455) | 4.43 (1.474) | NA (NA) — Results not reported for this group.

23. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2 (SF-36v2), Acute Components: Physical Functioning Domain
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. An additional item measures health transition. The 8 health domains are aggregated into two summary scores known as the PCS score and the MCS score. Norm-based domain scores, PCS and MCS scores are used in the analyses; each of which has a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher physical functioning domain score represents better physical functioning.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103,104, NA, NA, 103) | 2.43 (0.768) | 3.89 (0.776) | 2.81 (0.787) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 1.10 (0.840)
  Month 3 (n=102, 103,101, NA, NA, 102) | 5.17 (0.846) | 5.23 (0.848) | 5.22 (0.862) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 2.06 (0.910)
  Month 6 (n=100, 100, 99, 48, 48, NA) | 7.02 (0.897) | 6.15 (0.900) | 6.36 (0.912) | 5.22 (1.276) | 5.22 (1.291) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | 7.43 (0.902) | 6.67 (0.909) | 7.01 (0.921) | 5.69 (1.285) | 6.25 (1.306) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | 7.67 (0.899) | 7.11 (0.903) | 6.81 (0.917) | 6.49 (1.292) | 4.77 (1.308) | NA (NA) — Results were not reported for this group.

24. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2 (SF-36v2), Acute Components: Role-Physical Domain
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. An additional item measures health transition. The 8 health domains are aggregated into two summary scores known as the PCS score and the MCS score. Norm-based domain scores, PCS and MCS scores are used in the analyses; each of which has a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher role-physical domain score represents better role-physical functioning.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103,104, NA, NA, 103) | 4.05 (0.751) | 3.72 (0.759) | 4.09 (0.770) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 1.98 (0.820)
  Month 3 (n=102, 103, 100, NA, NA, 102) | 4.45 (0.801) | 4.79 (0.803) | 5.21 (0.820) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 3.63 (0.862)
  Month 6 (n=100, 100, 99, 48, 48, NA) | 6.02 (0.824) | 5.21 (0.828) | 5.48 (0.840) | 4.97 (1.172) | 5.03 (1.185) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | 6.24 (0.853) | 6.56 (0.861) | 5.79 (0.872) | 4.68 (1.217) | 6.70 (1.234) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | 6.21 (0.888) | 7.11 (0.892) | 6.37 (0.906) | 2.98 (1.279) | 5.03 (1.291) | NA (NA) — Results were not reported for this group.

25. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2 (SF-36v2), Acute Components: Bodily Pain Domain
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. An additional item measures health transition. The 8 health domains are aggregated into two summary scores known as the PCS score and the MCS score. Norm-based domain scores, PCS and MCS scores are used in the analyses; each of which has a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher bodily pain domain score represents less bodily pain.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103,104, NA, NA, 103) | 5.53 (0.777) | 7.16 (0.786) | 6.42 (0.802) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 3.44 (0.851)
  Month 3 (n=102, 103, 101, NA, NA, 102) | 7.75 (0.838) | 8.05 (0.840) | 7.52 (0.859) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 3.77 (0.903)
  Month 6 (n=100, 100, 99, 48, 48, NA) | 7.76 (0.985) | 10.65 (0.989) | 7.76 (1.004) | 8.55 (1.405) | 8.98 (1.425) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | 9.03 (0.953) | 10.13 (0.960) | 8.59 (0.977) | 8.46 (1.362) | 10.81 (1.389) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 43, NA) | 9.15 (0.961) | 11.38 (0.965) | 9.18 (0.984) | 8.59 (1.384) | 8.61 (1.413) | NA (NA) — Results were not reported for this group.

26. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2 (SF-36v2), Acute Components: General Health Domain
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. An additional item measures health transition. The 8 health domains are aggregated into two summary scores known as the PCS score and the MCS score. Norm-based domain scores, PCS and MCS scores are used in the analyses; each of which has a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher general health domain score represents better general health perceptions.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103,104, NA, NA, 103) | 3.29 (0.610) | 3.87 (0.616) | 1.96 (0.625) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 2.15 (0.666)
  Month 3 (n=102, 103,101, NA, NA, 102 ) | 4.09 (0.700) | 3.95 (0.701) | 4.73 (0.713) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 2.64 (0.748)
  Month 6 (n=100, 100, 99, 48, 48, NA) | 5.96 (0.720) | 4.12 (0.722) | 4.81 (0.733) | 4.39 (1.022) | 3.92 (1.033) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | 5.93 (0.773) | 5.18 (0.778) | 4.09 (0.788) | 4.72 (1.102) | 4.85 (1.117) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | 5.70 (0.811) | 4.63 (0.815) | 4.21 (0.825) | 4.50 (1.164) | 4.12 (1.175) | NA (NA) — Results were not reported for this group.

27. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2 (SF-36v2), Acute Components: Vitality Domain
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. An additional item measures health transition. The 8 health domains are aggregated into two summary scores known as the PCS score and the MCS score. Norm-based domain scores, PCS and MCS scores are used in the analyses; each of which has a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher vitality domain score represents better vitality.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103,104, NA, NA, 103) | 3.64 (0.802) | 4.59 (0.806) | 2.42 (0.826) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 2.16 (0.877)
  Month 3 (n=102, 103, 101, NA, NA, 102) | 5.50 (0.889) | 5.90 (0.887) | 4.93 (0.909) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 3.05 (0.954)
  Month 6 (n=100, 100, 99, 48, 48, NA) | 6.81 (0.969) | 7.41 (0.970) | 5.05 (0.989) | 5.34 (1.378) | 4.62 (1.394) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | 6.09 (1.017) | 7.82 (1.023) | 5.27 (1.041) | 6.61 (1.451) | 6.39 (1.472) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | 7.01 (1.022) | 7.02 (1.024) | 5.12 (1.043) | 5.62 (1.465) | 5.15 (1.481) | NA (NA) — Results were not reported for this group.

28. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2 (SF-36v2), Acute Components: Social Functioning Domain
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. An additional item measures health transition. The 8 health domains are aggregated into two summary scores known as the PCS score and the MCS score. Norm-based domain scores, PCS and MCS scores are used in the analyses; each of which has a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher social functioning domain score represents better social functioning.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable. n=number pf participants evaluable at each visit.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103,104, NA, NA, 103) | 4.51 (0.827) | 4.46 (0.838) | 3.34 (0.852) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 2.96 (0.901)
  Month 3 (n=102, 103, 101, NA, NA, 102) | 5.95 (0.897) | 5.22 (0.898) | 5.26 (0.918) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 3.63 (0.961)
  Month 6 (n=100, 100, 99, 48, 48, NA) | 6.97 (0.955) | 7.08 (0.959) | 7.10 (0.975) | 5.44 (1.362) | 6.05 (1.373) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | 7.66 (0.947) | 7.74 (0.957) | 5.69 (0.972) | 5.95 (1.355) | 8.93 (1.373) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | 6.13 (0.989) | 8.42 (0.995) | 6.32 (1.012) | 6.19 (1.427) | 6.41 (1.445) | NA (NA) — Results were not reported for this group.

29. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2 (SF-36v2), Acute Components: Role-Emotional Domain
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. An additional item measures health transition. The 8 health domains are aggregated into two summary scores known as the PCS score and the MCS score. Norm-based domain scores, PCS and MCS scores are used in the analyses; each of which has a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher role-emotional domain score represents better role-emotional functioning.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103,104, NA, NA, 103) | 4.77 (0.960) | 3.87 (0.971) | 2.93 (0.991) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | 4.52 (1.042)
  Month 3 (n=102, 103, 100, NA, NA, 102) | 4.21 (1.010) | 4.82 (1.011) | 3.35 (1.040) | NA (NA) — Results not reported for this group. | NA (NA) — Results not reported for this group. | 3.68 (1.083)
  Month 6 (n=100, 100, 98, 48, 48, NA) | 5.67 (1.024) | 4.68 (1.027) | 4.77 (1.051) | 6.34 (1.458) | 4.56 (1.473) | NA (NA) — Results not reported for this group.
  Month 9 (n=99, 97, 95, 47, 46, NA) | 5.13 (1.021) | 6.13 (1.030) | 4.87 (1.052) | 5.89 (1.456) | 6.52 (1.478) | NA (NA) — Results not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | 5.15 (1.048) | 6.73 (1.053) | 6.03 (1.075) | 4.77 (1.509) | 4.94 (1.525) | NA (NA) — Results not reported for this group.

30. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2 (SF-36v2), Acute Components: Mental Health Domain
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. An additional item measures health transition. The 8 health domains are aggregated into two summary scores known as the PCS score and the MCS score. Norm-based domain scores, PCS and MCS scores are used in the analyses; each of which has a population mean of 50 with a SD of 10 points, and ranges from minus infinity to plus infinity. A higher mental health domain score represents better mental health functioning.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103, 104, NA, NA, 103) | 3.32 (0.867) | 3.87 (0.874) | 2.79 (0.895) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 1.57 (0.952)
  Month 3 (n=102, 103, 101, NA, NA, 102) | 4.45 (0.934) | 4.23 (0.932) | 3.95 (0.956) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 2.62 (1.009)
  Month 6 (n=100, 100, 99, 48, 48, NA) | 6.11 (0.951) | 6.38 (0.953) | 5.35 (0.974) | 3.70 (1.354) | 3.41 (1.372) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | 5.79 (1.022) | 6.43 (1.028) | 4.62 (1.048) | 3.57 (1.461) | 5.45 (1.483) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | 5.86 (1.019) | 6.58 (1.022) | 5.86 (1.044) | 4.72 (1.467) | 4.48 (1.483) | NA (NA) — Results were not reported for this group.

31. Secondary Outcome: Change From Baseline in Score on EuroQol-5 Dimension Health State Profile (EQ-5D) and Change in Patient's Self-rated Health on a Vertical Visual Analogue Scale (VAS) Recorded on the EQ-5D Questionnaire (EQ-VAS): Mobility
Description: The EQ-5D is a descriptive system of health-related quality of life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take 1 of 3 responses. The responses record 3 levels of severity (no problems [1], some or moderate problems [2], or extreme problems [3]) within a particular EQ-5D dimension. Standard vertical 0 to 100 mm visual analogue scale (similar to a thermometer) for recording an individual's rating for their current health-related quality of life state, with a higher value representing better health status.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103, 104, NA, NA, 103) | -0.07 (0.042) | -0.19 (0.043) | -0.15 (0.043) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -0.10 (0.046)
  Month 3 (n=101, 103, 101, NA, NA, 102) | -0.28 (0.047) | -0.27 (0.047) | -0.29 (0.048) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -0.11 (0.050)
  Month 6 (n=100, 100, 99, 48, 48, NA) | -0.3 (0.05) | -0.3 (0.05) | -0.2 (0.05) | -0.3 (0.07) | -0.2 (0.07) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | -0.3 (0.05) | -0.3 (0.05) | -0.3 (0.05) | -0.3 (0.07) | -0.3 (0.07) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44,44, NA) | -0.3 (0.05) | -0.3 (0.05) | -0.3 (0.05) | -0.4 (0.07) | -0.3 (0.07) | NA (NA) — Results were not reported for this group.

32. Secondary Outcome: Change From Baseline in Score on EuroQol-5 Dimension Health State Profile (EQ-5D) and Change in Patient's Self-rated Health on a Vertical Visual Analogue Scale (VAS) Recorded on the EQ-5D Questionnaire (EQ-VAS): Self-care
Description: as for outcome 31
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 103 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 102, 104, NA, NA, 103) | -0.11 (0.046) | -0.16 (0.047) | -0.16 (0.047) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -0.09 (0.050)
  Month 3 (n=101, 102, 101, NA, NA, 102) | -0.19 (0.047) | -0.11 (0.047) | -0.18 (0.048) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -0.12 (0.051)
  Month 6 (n=100, 99, 99, 48, 48, NA) | -0.2 (0.04) | -0.3 (0.05) | -0.2 (0.05) | -0.2 (0.06) | -0.3 (0.06) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | -0.2 (0.05) | -0.2 (0.05) | -0.3 (0.05) | -0.2 (0.06) | -0.3 (0.07) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | -0.2 (0.05) | -0.3 (0.05) | -0.3 (0.05) | -0.3 (0.07) | -0.2 (0.07) | NA (NA) — Results were not reported for this group.

33. Secondary Outcome: Change From Baseline in Score on EuroQol-5 Dimension Health State Profile (EQ-5D) and Change in Patient's Self-rated Health on a Vertical Visual Analogue Scale (VAS) Recorded on the EQ-5D Questionnaire (EQ-VAS): Usual Activities
Description: as for outcome 31
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 103 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 102, 104, NA, NA, 103) | -0.17 (0.043) | -0.19 (0.043) | -0.21 (0.044) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -0.06 (0.047)
  Month 3 (n=101, 102, 101, NA, NA, 102) | -0.24 (0.049) | -0.29 (0.049) | -0.29 (0.049) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -0.17 (0.052)
  Month 6 (n=100, 99, 99, 48, 47, NA) | -0.3 (0.05) | -0.3 (0.05) | -0.4 (0.05) | -0.3 (0.07) | -0.3 (0.07) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | -0.3 (0.05) | -0.4 (0.05) | -0.4 (0.05) | -0.3 (0.07) | -0.4 (0.07) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | -0.3 (0.05) | -0.4 (0.05) | -0.4 (0.05) | -0.3 (0.07) | -0.3 (0.07) | NA (NA) — Results were not reported for this group.

34. Secondary Outcome: Change From Baseline in Score on EuroQol-5 Dimension Health State Profile (EQ-5D) and Change in Patient's Self-rated Health on a Vertical Visual Analogue Scale (VAS) Recorded on the EQ-5D Questionnaire (EQ-VAS): Pain/Discomfort
Description: as for outcome 31
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103, 104, NA, NA, 103) | -0.14 (0.039) | -0.25 (0.040) | -0.19 (0.040) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -0.08 (0.043)
  Month 3 (n=101, 103, 101, NA, NA, 102) | -0.25 (0.044) | -0.27 (0.044) | -0.28 (0.045) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -0.08 (0.047)
  Month 6 (n=100, 100, 99, 48, 48, NA) | -0.3 (0.05) | -0.4 (0.05) | -0.3 (0.05) | -0.3 (0.07) | -0.4 (0.07) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | -0.3 (0.05) | -0.3 (0.05) | -0.3 (0.05) | -0.4 (0.07) | -0.4 (0.07) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | -0.3 (0.05) | -0.4 (0.05) | -0.3 (0.05) | -0.2 (0.07) | -0.3 (0.07) | NA (NA) — Results were not reported for this group.

35. Secondary Outcome: Change From Baseline in Score on EuroQol-5 Dimension Health State Profile (EQ-5D) and Change in Patient's Self-rated Health on a Vertical Visual Analogue Scale (VAS) Recorded on the EQ-5D Questionnaire (EQ-VAS): Anxiety/Depression
Description: as for outcome 31
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103, 104, NA, NA, 103) | -0.25 (0.051) | -0.22 (0.052) | -0.27 (0.053) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -0.21 (0.056)
  Month 3 (n=101, 103, 100, NA, NA, 102) | -0.25 (0.055) | -0.17 (0.055) | -0.32 (0.056) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -0.21 (0.059)
  Month 6 (n=100, 100, 99, 48, 48, NA) | -0.3 (0.05) | -0.3 (0.05) | -0.3 (0.05) | -0.3 (0.08) | -0.2 (0.08) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | -0.3 (0.05) | -0.4 (0.05) | -0.4 (0.06) | -0.2 (0.08) | -0.3 (0.08) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | -0.3 (0.05) | -0.4 (0.05) | -0.4 (0.06) | -0.2 (0.08) | -0.3 (0.08) | NA (NA) — Results were not reported for this group.

36. Secondary Outcome: Change From Baseline in Score on EuroQol-5 Dimension Health State Profile (EQ-5D) and Change in Patient's Self-rated Health on a Vertical Visual Analogue Scale (VAS) Recorded on the EQ-5D Questionnaire (EQ-VAS): Patient's Health State Today
Description: The EQ-5D is a descriptive system of health-related quality of life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take 1 of 3 responses. The responses record 3 levels of severity (no problems [1], some or moderate problems [2], or extreme problems [3]) within a particular EQ-5D dimension. Standard vertical 0 (worst imaginable health state) to 100 mm (best imaginable health state) visual analogue scale (similar to a thermometer) for recording an individual's rating for their current health-related quality of life state; higher scores indicate a better health state, with a higher value representing better health status.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
mm
  Month 1 (n=105, 103, 104, NA, NA, 103) | 10.75 (1.859) | 10.81 (1.880) | 10.27 (1.917) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 6.59 (2.027)
  Month 3 (n=101, 103, 101, NA, NA, 101) | 14.00 (2.100) | 15.83 (2.092) | 13.10 (2.138) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 6.37 (2.242)
  Month 6 (n=100, 100, 99, 48, 48, NA) | 19.5 (2.08) | 15.7 (2.09) | 15.5 (2.12) | 14.7 (2.97) | 16.6 (3.00) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | 19.2 (2.21) | 15.9 (2.23) | 18.2 (2.26) | 12.8 (3.16) | 21.5 (3.21) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | 20.7 (2.09) | 19.8 (2.09) | 16.5 (2.14) | 16.0 (3.02) | 19.8 (3.05) | NA (NA) — Results were not reported for this group.

37. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Scores: Total Score
Description: FACIT-F is a 13-item questionnaire, with each item scored on a 5-point scale ranging from 0 (not at all) to 4 (very much). Three endpoints are derived: change in FACIT-F total score, change in FACIT-F experience domain score, and change in FACIT-F impact domain score. FACIT-F total score (range 0 to 52) is calculated by summing the 13 items. FACIT-F experience domain score (range 0-20) is calculated by summing 5 items : I feel fatigued, I feel weak all over, I feel listless ("washed out"), I feel tired, and I have energy, while FACIT-F impact domain score (range 0-32) is calculated by summing the remaining 8 items. All responses are added with equal weight to obtain the total score. Higher scores represent better fatigue status.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103, 104, NA, NA, 103) | 5.2 (0.77) | 4.4 (0.78) | 4.2 (0.79) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 2.7 (0.84)
  Month 3 (102, 102, 101, NA, NA, 102) | 7.0 (0.85) | 6.0 (0.85) | 6.0 (0.87) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 3.3 (0.91)
  Month 6 (n=100, 100, 99,48, 48, NA) | 7.9 (0.89) | 8.0 (0.89) | 6.5 (0.91) | 6.5 (1.26) | 7.2 (1.28) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | 7.9 (0.92) | 7.4 (0.92) | 6.5 (0.94) | 5.5 (1.31) | 8.4 (1.33) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | 8.5 (0.95) | 8.4 (0.95) | 6.9 (0.97) | 5.7 (1.36) | 7.6 (1.38) | NA (NA) — Results were not reported for this group.

38. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Scores: Experience Domain Score
Description: FACIT-F is a 13-item questionnaire, with each item score ranging from 0 to 4. Three endpoints are derived: change in FACIT-F total score, change in FACIT-F experience domain score, and change in FACIT-F impact domain score. FACIT-F total score (range 0-52) is calculated by summing the 13 items. FACIT-F experience domain score (range 0-20) is calculated by summing 5 items : I feel fatigued, I feel weak all over, I feel listless ("washed out"), I feel tired, and I have energy, while FACIT-F impact domain score (range 0-32) is calculated by summing the remaining 8 items. All responses are added with equal weight to obtain the total score. Higher scores represent better (less) fatigue experience.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103, 104, NA, NA, 103) | 2.4 (0.35) | 2.1 (0.35) | 2.1 (0.36) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 1.2 (0.38)
  Month 3 (n=102, 102, 101, NA, NA, 102) | 3.3 (0.38) | 2.8 (0.38) | 2.9 (0.39) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 1.6 (0.41)
  Month 6 (n=100, 100, 99,48, 48, NA) | 3.6 (0.40) | 3.3 (0.40) | 3.2 (0.41) | 3.0 (0.57) | 3.3 (0.58) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | 3.6 (0.42) | 3.3 (0.42) | 3.3 (0.43) | 2.7 (0.59) | 3.9 (0.60) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | 3.9 (0.44) | 3.7 (0.44) | 3.2 (0.45) | 2.7 (0.63) | 3.4 (0.63) | NA (NA) — Results were not reported for this group.

39. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Scores: Impact Domain Score
Description: FACIT-F is a 13-item questionnaire, with each item score ranging from 0 to 4. Three endpoints are derived: change in FACIT-F total score, change in FACIT-F experience domain score, and change in FACIT-F impact domain score. FACIT-F total score (range 0-52) is calculated by summing the 13 items. FACIT-F experience domain score (range 0-20) is calculated by summing 5 items : I feel fatigued, I feel weak all over, I feel listless ("washed out"), I feel tired, and I have energy, while FACIT-F impact domain score (range 0-32) is calculated by summing the remaining 8 items. All responses are added with equal weight to obtain the total score. Higher scores represent better (less) fatigue impact on daily functioning.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 106 | 104 | 106 | 52 | 52 | 104
Units on a scale
  Month 1 (n=105, 103, 104, NA, NA, 103) | 2.9 (0.47) | 2.3 (0.48) | 2.1 (0.49) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 1.5 (0.52)
  Month 3 (n=102, 102, 101, NA, NA, 102) | 3.8 (0.52) | 3.2 (0.52) | 3.2 (0.53) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | 1.8 (0.56)
  Month 6 (n=100, 100, 99,48, 48, NA) | 4.3 (0.53) | 4.7 (0.53) | 3.4 (0.54) | 3.5 (0.75) | 4.0 (0.76) | NA (NA) — Results were not reported for this group.
  Month 9 (n=99, 97, 96, 47, 46, NA) | 4.3 (0.55) | 4.1 (0.55) | 3.3 (0.56) | 2.8 (0.78) | 4.6 (0.80) | NA (NA) — Results were not reported for this group.
  Month 12 (n=96, 96, 94, 44, 44, NA) | 4.6 (0.57) | 4.7 (0.57) | 3.7 (0.58) | 2.9 (0.82) | 4.3 (0.82) | NA (NA) — Results were not reported for this group.

40. Secondary Outcome: Change From Baseline in Scores Evaluating Spondylitis Using the Bath Anklyosing Spondylitis Disease Activity Index (BASDAI)
Description: BASDAI is a validated self-assessment tool used to determine disease activity in participants with ankylosing spondylitis. Utilizing a visual analog scale of 0-100mm (0=none and 100=very severe) participants answer 6 questions measuring discomfort, pain, and fatigue. The final BASDAI score averages the individual assessments for a final score ranging 0-10cm, with higher scores representing more severe ankylosing spondylitis disease activity.
Time Frame: From Baseline to Months 1, 3, 6, 9, and 12
Population: All participants who were randomized, received at least 1 dose of study drug with presence of spondylitis at screening and baseline BASDAI score>0 cm and were evaluable. n=number of participants evaluable at each visit.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 24 | 21 | 10 | 10 | 12 | 22
cm
  Month 1 (n=24, 21, 10, NA, NA, 22) | -1.23 (0.537) | -1.60 (0.508) | -2.30 (0.673) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -1.27 (0.581)
  Month 3 (n=24, 21, 10, NA, NA, 22) | -1.83 (0.579) | -2.78 (0.559) | -2.93 (0.753) | NA (NA) — Results were not reported for this group. | NA (NA) — Results were not reported for this group. | -1.60 (0.624)
  Month 6 (n=23, 21, 10, 9, 11, NA) | -2.24 (0.580) | -2.35 (0.560) | -3.58 (0.758) | -2.85 (0.778) | -3.31 (0.744) | NA (NA) — Results were not reported for this group.
  Month 9 (n=23, 20, 10, 9, 9, NA) | -2.06 (0.575) | -2.71 (0.558) | 2.66 (0.747) | -3.00 (0.770) | -3.35 (0.761) | NA (NA) — Results were not reported for this group.
  Month 12 (n=23, 19, 10, 9, 9, NA) | -2.50 (0.594) | -3.30 (0.587) | -2.42 (0.779) | -2.31 (0.808) | -2.67 (0.806) | NA (NA) — Results were not reported for this group.

ADVERSE EVENTS:
Arm/Group | Tofacitinib, 5 mg, Twice Daily | Tofacitinib, 10 mg, Twice Daily | Adalimumab, 40 mg, Every 2 Weeks | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily
Serious Adverse Events (participants affected / at risk) | 8/107 | 4/104 | 9/106 | 3/52 | 4/53
Other Adverse Events (participants affected / at risk) | 31/107 | 43/104 | 43/106 | 15/52 | 22/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib, 5 mg, Twice Daily (N=107) | Tofacitinib, 10 mg, Twice Daily (N=104) | Adalimumab, 40 mg, Every 2 Weeks (N=106) | Placebo/Tofacitinib, 5 mg, Twice Daily (N=52) | Placebo/Tofacitinib, 10 mg, Twice Daily (N=53)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyoderma streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib, 5 mg, Twice Daily (N=107) | Tofacitinib, 10 mg, Twice Daily (N=104) | Adalimumab, 40 mg, Every 2 Weeks (N=106) | Placebo/Tofacitinib, 5 mg, Twice Daily (N=52) | Placebo/Tofacitinib, 10 mg, Twice Daily (N=53)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 3
Nausea (Gastrointestinal disorders) | 3 | 4 | 6 | 0 | 1
Nasopharyngitis (Infections and infestations) | 8 | 12 | 11 | 4 | 4
Pharyngitis (Infections and infestations) | 5 | 6 | 7 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 10 | 11 | 8 | 5 | 5
Urinary tract infection (Infections and infestations) | 2 | 4 | 4 | 1 | 4
Alanine aminotransferase increased (Investigations) | 3 | 3 | 8 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 7 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 5 | 5 | 3 | 1 | 5
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 3 | 0
Headache (Nervous system disorders) | 5 | 11 | 7 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.